CLINICAL TRIAL: NCT07027033
Title: Nutritional Oleic Acid Modulation of adIpose Cholesterol Metabolism in Patients Living With Obesity
Acronym: NAMICO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RC24_0626; 2024-A02770-47 (Registry Identifier: ID RCB)
Record Dates: First submitted 2025-05-16; First posted 2025-06-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Visceral Adipose Tissue; White Adipose Tissue Inflammation; Subcutaneous Adipose Tissue
Keywords: obesity; visceral adipose tissue; adipocyte dysfunction; oleic acid; cholesterol esterification
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: NAMICO is a physio-pathologic, monocentric, controlled , blinded, randomized trial
Who Masked: Care Provider, Investigator
Masking Description: Oil bottles will be numbered in accordance with a correspondence list generated electronically by the datamanager (blinding procedure for participant, investigator and their team).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oleic acid group (Experimental): Female patients undergoing bariatric surgery will be asked to adjust their oleic acid intake through a nutritional, non-pharmacological intervention. This involves the consumption of 40 ml of sunflower oil rich in oleic acid. Of this amount, 30 mL consumed in two portions: one tablespoon (approximately 15 mL) in the morning or at lunch time, and another in the evening. The remaining 10 mL will be used as a substitute for usual dietary fats. This diet will be followed for approximately 13 weeks prior to bariatric surgery.
  Interventions: Other: acid-rich sunflower oil oleic acid
- Conventional oil group (control group) (Placebo Comparator): Female patients undergoing bariatric surgery will be asked to adjust their dietary intake of sunflower oil. This involves the consumption of 40 ml of sunflower (composition of the sunflow oil only differs fatty acid composition). Of this amount, 30 mL consumed in two portions: one tablespoon (approximately 15 mL) in the morning or at lunch time, and another in the evening. The remaining 10 mL will be used as a substitute for usual dietary fats. This diet will be followed for approximately 13 weeks prior to bariatric surgery.
  Interventions: Other: conventional sunflower oil

INTERVENTIONS:
Other: acid-rich sunflower oil oleic acid — Nutritional intervention for 13 weeks ± 2 weeks, including 40 millilitres of sunflower oil rich in oleic acid
  Arms: Oleic acid group
Other: conventional sunflower oil — Nutritional intervention for 13 weeks ± 2 weeks, including 40 millilitres of conventional sunflower oil
  Arms: Conventional oil group (control group)

SUMMARY:
Disruption of white adipose tissue (WAT) homeostasis during obesity is central to the development of associated cardiometabolic complications. Dietary supplementation with oleic acid in obese patients can limit these complications. Experimental data, obtained in preclinical models, suggest that the beneficial effects of oleic acid may protect the TAB by increasing cholesterol esterification. The NAMICO study aims to test this hypothesis using TAB biopsies collected from obese patients undergoing bariatric surgery who had previously undergone dietary enrichment with either a conventional oil or an oil rich in oleic acid.

ELIGIBILITY:
Inclusion Criteria:

* • Individual who has given informed consent.

  * Female adult aged between 18 and 60 years (included).
  * Patient with obesity at inclusion, meeting the HAS criteria for bariatric surgery eligibility: BMI ≥ 35 kg/m² associated with a comorbidity or BMI > 40 kg/m².
  * European origin: For this pilot study, we need to reduce variability factors and focus the research on women of European descent only (having both parents identified by the patient as of European origin).
  * Effective contraception if sexually active, or abstinence, or menopause (criterion required for bariatric surgery).
  * Presenting at inclusion with at least two clinical criteria of insulin resistance according to the definition of the International Diabetes Federation (IDF):

    * Dysglycemia (fasting glucose ≥ 100 mg/dL, glucose intolerance, or type 2 diabetes).
    * Hypertension (≥ 130/85 mm Hg).
    * Low HDL-cholesterol (< 50 mg/dL).
    * Elevated triglycerides (≥ 150 mg/dL).
  * Affiliated with a social security system or a beneficiary of such a system.
  * Bariatric surgery performed at Nantes University Hospital (CHU de Nantes).

Exclusion Criteria:

* • Modification of diabetes treatment within the past month.

  * Ongoing or planned insulin therapy before bariatric surgery.
  * Modification of lipid-lowering treatment within the past three months.
  * Systemic corticosteroid therapy.
  * Antiviral therapy (HIV).
  * Dietary supplementation affecting lipid metabolism, including proactive margarine, Danacol, polyunsaturated fatty acid supplementation, or any other substance identified by the investigator.
  * Exocrine pancreatic insufficiency.
  * Pregnancy or breastfeeding.
  * History of organ transplantation.
  * Individual deprived of liberty or under legal protection (guardianship or trusteeship).
  * Any clinical condition in which the investigator considers that inclusion in the study may harm the patient's health or compromise the proper conduct of the study.
  * Participation in other clinical trials, except for non-interventional studies and research on surgical techniques or postoperative strategies.

    * Type I, monogenic or secondary diabetes.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of consuming oleic acid-rich sunflower oil versus conventional sunflower oil on cholesterol esterification within visceral white adipose tissue. | 13 weeks +/- 2 week
  The primary endpoint of the study is to compare the cholesterol esterification rates in adipocytes between the two experimental groups. This is measured by the ratio of esterified cholesterol (EC) to free cholesterol (FC), expressed as a percentage, determined from samples of visceral adipose tissue collected perioperatively after 13 weeks (± 2 week) of the nutritional supplementation under investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Marie De Montrichard, PH, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France, France

IPD SHARING:
Plan to Share IPD: No